CLINICAL TRIAL: NCT03778320
Title: A Randomized Single Dose Crossover Comparison of the Safety, Tolerability, and Pharmacokinetic Profile of CTP-692 Versus D-Serine
Brief Title: A Study to Compare the Safety, Tolerability, and Pharmacokinetics of CTP-692 Versus D-serine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP692.1001
Record Dates: First submitted 2018-12-13; First posted 2018-12-19 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTP-692 (Experimental)
  Interventions: Drug: CTP-692
- D-Serine (Active Comparator)
  Interventions: Drug: D-Serine

INTERVENTIONS:
Drug: CTP-692 — Single oral dose
  Arms: CTP-692
Drug: D-Serine — Single oral dose
  Arms: D-Serine

SUMMARY:
This study will assess the safety, tolerability and pharmacokinetic (PK) profile of CTP-692 vs D serine.

ELIGIBILITY:
Inclusion Criteria:

* Must give written and informed consent and any authorizations required by local law.
* Must have a body mass index (BMI) between 18 kg/m2 and 32 kg/m2, inclusive

Exclusion Criteria:

* Screening laboratory measurements outside the normal range associated with potential risk for the treatment under investigation at screening and/or prior to the first dose of study drug
* Positive blood screen for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen or hepatitis C virus antibody
* History of clinically significant central nervous system (e.g., seizures), cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal (GI) conditions
* Positive drug or alcohol test at screening or prior to the first dose of study drug

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2018-12-23 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
The number of AEs in participants as a measure of safety and tolerability. | 7 days
Measurement of CTP-692 exposure in plasma | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Emily McIntyre, Study Director — Concert Pharmaceuticals, Inc.
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No